CLINICAL TRIAL: NCT03631745
Title: Delivering Church-based Interventions to Reduce Stigma and Mental Health Treatment Disparities Among Latinos
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Collaborators: National Alliance on Mental Illness California (Unknown)
Responsible Party: Principal Investigator, Eunice Wong, Senior Behavioral Scientist, RAND
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: R01MD012638 (NIH)
Record Dates: First submitted 2018-08-02; First posted 2018-08-15 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Help-Seeking Behavior; Stigma, Social
Keywords: mental health literacy; stigma; help-seeking; Latino; faith-based; religious congregations; contact-based interventions
MeSH Terms: conditions — Help-Seeking Behavior; Social Stigma

STUDY DESIGN:
Intervention Model Description: The National Alliance on Mental Illness (NAMI) of California has developed Mental Health 101, a suite of contact-based education programs tailored for culturally diverse populations including Latino populations. Another NAMI program, FaithNet, provides resources and training on how churches can shape norms and overcome shame and stigma related to mental illness and treatment. NAMI FaithNet also assists with facilitating linkages to mental health services from providing referrals to partner mental health agencies to forming multi-sector collaboratives of social service organizations, clergy, and mental health providers to create a more holistic, coordinated system of care. The multi-component, church-based, intervention will build on NAMI's existing resources, with tailoring for Latino church-based settings.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NAMI Mental Health 101 and NAMI FaithNet (Experimental): Mental Health 101 and FaithNet
  Interventions: Behavioral: NAMI Mental Health 101 and NAMI FaithNet
- Wait-list Control (No Intervention): After the 12-month follow-up, wait-list control churches will be provided with the opportunity to receive Mental Health 101 and NAMI FaithNet interventions.

INTERVENTIONS:
Behavioral: NAMI Mental Health 101 and NAMI FaithNet — Congregants of Intervention Churches will receive:
  1. NAMI Mental Health 101, a 60-90 minute, contact-based educational intervention
  2. NAMI FaithNet which consists of congregational support and training to cultivate supportive environments within faith communities for those with mental health conditions and their families.
  Arms: NAMI Mental Health 101 and NAMI FaithNet

SUMMARY:
This study is a cluster randomized controlled trial of a Latino church-based intervention in Los Angeles and Riverside Counties. This study aims to leverage the collective resources of Latino religious congregations and the National Alliance on Mental Illness to test the effectiveness of a multi-component intervention directed at reducing stigma, increasing mental health literacy, and improving access to mental health services.

DETAILED DESCRIPTION:
This study is a cluster randomized controlled trial of a Latino church-based intervention in Los Angeles and Riverside Counties. This study aims to leverage the collective resources of Latino religious congregations and the National Alliance on Mental Illness to test the effectiveness of a multi-component intervention directed at reducing stigma, increasing mental health literacy, and improving access to mental health services. A total of 12 churches (6 intervention and 6 wait-list control) will be enrolled in the study. Churches within each study site, the Riverside County parishes and the Archdiocese of Los Angeles, will be matched in pairs based on size and geography. Three matched pairs from each study site will be randomly selected and then randomly assigned within each pair to intervention or control. The planned study will involve 2400 participants (1200 intervention and 1200 control) who will be part of congregations that are randomly assigned to receive the church-based intervention immediately or a wait list control condition. Participants will be assessed at baseline, 6-month follow-up, and 12-month follow-up to evaluate intervention effects on mental health service use and potential mediators (i.e., mental health literacy, stigma).

ELIGIBILITY:
Inclusion Criteria:

* Congregant of selected intervention and control churches

Exclusion Criteria:

* Does not meet criteria above

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1713 (Actual)
Dates: Start 2020-02-09 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Mental Health Service Use | Mental Health Service Use between Baseline and 12-month Follow-up
  Change in mental health service use among participants in intervention churches versus those in control churches.
  Mental health service use will be measured with the following modified item from the California Health Interview Survey: "In the past 12 months have you seen a professional, such as a counselor, psychiatrist, or social worker for problems with your mental health, emotions, nerves, or your use of alcohol or drugs?"
  Response options are dichotomous (Yes/No).
  Tran LD, Ponce NA. Who Gets Needed Mental Health Care? Use of Mental Health Services among Adults with Mental Health Need in California. Calif J Health
  Promot. 2017;15(1):36-45. PubMed PMID: 28729814; PubMed Central PMCID:
  PMC5515380.

SECONDARY OUTCOMES:
Mental Illness Stigma | Mental Illness Stigma reduction between Baseline and 12-month Follow-up
  Change in stigma among participants in intervention churches versus those in control churches. Personal stigma will be assessed with social distance measures, one of the most widely used indicators of stigma. Social distance is assessed by asking respondents to rate their degree of willingness to interact with someone with a mental illness in various interpersonal situations (e.g., work closely on a job; live next door; spend an evening socializing; marry into the family; as a friend).
  Jorm AF, Oh E. Desire for social distance from people with mental disorders. The Australian and New Zealand journal of psychiatry. 2009;43(3):183-200.

CONTACTS AND LOCATIONS:
Overall Officials: Eunice C Wong, Principal Investigator — RAND
Locations (1):
- RAND, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wong EC, Martinez MO, Han B, Seelam R, Derose KP. Cluster-Randomized Trial of a Multilevel Parish-Based Intervention to Improve Mental Health Literacy and Reduce Stigma in Hispanic Communities. Res Sq [Preprint]. 2025 Oct 26:rs.3.rs-7017764. doi: 10.21203/rs.3.rs-7017764/v1. PMID 41282142

DOCUMENTS (1):
  • Informed Consent Form (2020-12-01): https://cdn.clinicaltrials.gov/large-docs/45/NCT03631745/ICF_000.pdf